CLINICAL TRIAL: NCT01292824
Title: Phase I Study of Hepatitis C Virus (HCV) Entry Inhibitor (ITX 5061) in Liver Transplant Recipients With HCV Infection
Brief Title: Pilot Study of Hepatitis C Virus Entry Inhibitor (ITX 5061) in Liver Transplant Recipients
Acronym: ITX5061
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: University Hospital Birmingham (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_10-104; 2010-020358-32 (EudraCT Number)
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Hepatitis C; Evidence of Liver Transplantation
Keywords: Hepatitis C virus; Entry; Scavenger receptor-BI; High density lipoprotein; Liver transplantation
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard liver transplant care (No Intervention): Liver Transplantation as per Standard of Care
- ITX 5061 (Experimental): Liver Transplantation as per Standard of Care + ITX5061
  Interventions: Drug: ITX 5061

INTERVENTIONS:
Drug: ITX 5061 — ITX 5061 (150mg) pre-transplant, immediately post-transplant and daily thereafter for 1 week.
  Arms: ITX 5061

SUMMARY:
This is a phase I pilot study to determine the safety and preliminary efficacy of a novel hepatitis C virus (HCV) entry inhibitor (ITX 5061) in patients with HCV infection undergoing liver transplantation.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection is common and treatment options at present are limited. Recurrence of HCV infection after liver transplantation is inevitable and disease progression is rapid when compared with disease in the non-transplanted liver.

Studies of ITX 5061 in vitro have shown it to be a potent inhibitor of HCV entry into hepatocytes, through blocking the interaction of the virus with scavenger receptor BI suggesting it may reduce graft re-infection rates after liver transplant.

There are no studies of treatments to block host receptors for HCV and the investigators hypothesize that ITX 5061 will modulate HCV kinetics in the early phase post liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, ≤ 65 years old
* Plasma HCV RNA positive at time of listing for liver transplantation
* Accepted for liver transplantation for any of:
* End-stage liver disease due to HCV infection
* End-stage liver disease due to HCV infection and alcohol related liver disease (ALD)
* HCC due to HCV

Exclusion Criteria:

* Refusal or inability to give informed consent
* Viral co-infection with either hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* Pregnancy or breastfeeding
* Women, of child-bearing potential, who are not willing to practice effective contraception
* Men, sexually active with women of child-bearing potential, who are not willing to practice effective contraception
* Any situation that in the Investigator's opinion may interfere with optimal study participation
* Participation in any clinical study of an investigational agent within 30 days of recruitment
* Transplantation with a donor organ from a HCV positive individual

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To determine the safety of ITX 5061 in liver transplant recipients | 90 days
  Safety will be assessed by determination of the frequency of:
  * perioperative events: including transfusion requirements and vasopressor requirements
  * post-operative events: including primary graft non-function, hepatic artery thrombosis, acute cellular rejection and infective complications

SECONDARY OUTCOMES:
To determine whether treatment leads to an alteration in HCV RNA kinetics in the first week after liver transplantation | One week
  Hepatitis C virus titers will be measured at multiple times in the peri- and immediate post-operative period and kinetics assessed at 7 days after liver transplant.
To determine whether any change in early viral kinetics is sustained | 90 days
  Hepatitis C virus titers will be measured at multiple times in the post-operative period and kinetics assessed at 90 days after liver transplant.

CONTACTS AND LOCATIONS:
Overall Officials: David J Mutimer, FRCP, Principal Investigator — University of Birmingham
Locations (1):
- University Hospital Birmingham, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Background] Syder AJ, Lee H, Zeisel MB, Grove J, Soulier E, Macdonald J, Chow S, Chang J, Baumert TF, McKeating JA, McKelvy J, Wong-Staal F. Small molecule scavenger receptor BI antagonists are potent HCV entry inhibitors. J Hepatol. 2011 Jan;54(1):48-55. doi: 10.1016/j.jhep.2010.06.024. Epub 2010 Aug 21. PMID 20932595
- [Result] Rowe IA, Tully DC, Armstrong MJ, Parker R, Guo K, Barton D, Morse GD, Venuto CS, Ogilvie CB, Hedegaard DL, McKelvy JF, Wong-Staal F, Allen TM, Balfe P, McKeating JA, Mutimer DJ. Effect of scavenger receptor class B type I antagonist ITX5061 in patients with hepatitis C virus infection undergoing liver transplantation. Liver Transpl. 2016 Mar;22(3):287-97. doi: 10.1002/lt.24349. PMID 26437376